CLINICAL TRIAL: NCT00350142
Title: Phase II Study to Evaluate the Efficacy of Trilogy Stereotactic Radiosurgery for Pancreatic Cancer
Brief Title: Trilogy Stereotactic Body Radiotherapy for Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Koong (Other)
Responsible Party: Sponsor-Investigator, Albert Koong, Associate Professor of Radiation Oncology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANC0005; PANC0005 (Other: Stanford OnCore)
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2016-12

CONDITIONS: Pancreatic Cancer
Keywords: Stereotactic Body Radiotherapy (SBRT); pancreas cancer; locally advanced; local control; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery; Gemcitabine; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Body Radiotherapy (Experimental): Patients will have a 4D pancreatic protocol CT and a FDG PET scan scan, both for planning purposes. An SBRT treatment plan will be developed based on tumor geometry and location. All patients will receive a single fraction of 25 Gy dose of Stereotactic Body Radiotherapy on Trilogy Linear Accelerator, followed by weekly Gemcitabine.
  Interventions: Radiation: Stereotactic Body Radiotherapy; Drug: Gemcitabine; Other: 4D pancreatic protocol CT scan; Radiation: FDG PET scan

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — Stereotactic Body Radiotherapy will be performed using Trilogy Linear Accelerator
  Other Names: single fraction 25 Gy dose Stereotactic Body Radiotherapy
Drug: Gemcitabine — Weekly Gemcitabine will be administered at 1000mg/m2 over 100 minutes
  Other Names: Gemzar
Other: 4D pancreatic protocol CT scan — Patients will undergo this imaging procedure prior to treatment for planning purposes.
  Other Names: computerized tomography scan
Radiation: FDG PET scan — Patients will have this imaging procedure along with a CT scan to map the tumor and facilitate treatment planning.
  Other Names: Fluorodeoxyglucose (FDG)-positron emission tomography

SUMMARY:
This study will assess the efficacy of treating locally advanced pancreatic cancer using Stereotactic Body Radiotherapy (using Trilogy) and Gemcitabine

DETAILED DESCRIPTION:
In this study, we propose to combine stereotactic body radiotherapy (SBRT) with standard gemcitabine chemotherapy. We hypothesize that earlier administration of systemic chemotherapy may prolong the interval to distant progression and improve overall survival in these patients. In this study, we will treat pancreatic cancer patients with locally advanced disease with 3 weeks of gemcitabine, followed by Trilogy(TM) SBRT and additional gemcitabine. 30 patients will be accrued to this study at Stanford University Medical Center, the only site participating in this research study. Treatment on this protocol requires placement of 3-5 gold (99.9% pure) fiducials for targeting purposes. Four to 7 days after placement of the fiducials, patients will then undergo a 4D pancreatic protocol CT scan through the upper abdomen. In addition, an FDG PET scan is required for treatment planning purposes. This imaging set will be processed for radiosurgery, using a modified linac based radiation treatment planning system (EclipseTM). An SBRT treatment plan will be developed based on tumor geometry and location. All patients will receive a single fraction of 25 Gy prescribed to the isodose line that completely surrounds the gross pancreatic tumor volume (GTV) as defined by the contrast CT. Following SBRT, patients will be monitored clinically and radiographically.

ELIGIBILITY:
Inclusion Criteria:- Pancreatic tumors not to exceed 10 cm in greatest axial dimension

* Histologically confirmed malignancies of the pancreas
* Unresectable by CT criteria or exploratory laparotomy or laparoscopy
* Patients with metastatic disease may be treated if they are symptomatic from the primary tumor
* Performance status of 0, 1, or 2
* No chemotherapy two weeks prior or two weeks following radiosurgery

Exclusion Criteria:

* patients who have had prior radiotherapy to upper abdomen
* patients receiving any prior pancreatic cancer therapy
* children, pregnant, and breastfeeding women, and lab personnel are excluded
* uncontrolled intercurrent illnesses
* any concurrent malignancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Koong, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Stereotactic Body Radiotherapy: patients that received a single fraction of 25 Gy Stereotactic Body Radiotherapy followed by weekly Gemcitabine administered at 1000mg/m2 over 100 minutes.
  Patients will be followed at 4-6 weeks, 3 months, 6 months, 9 months and 1 year, in year 2 follow up will be every 4 months and in year 3 follow up will be every 6 months.
Period: Overall Study
Arm/Group | Stereotactic Body Radiotherapy
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- SBRT: 25 Gy single fraction dose using Trilogy linear accelerator
Arm/Group | SBRT
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 63 [45 to 85]
Gender [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Rate of Local Control
Description: The proportion of patients with local control where local control is defined as no recurrence or disease progression in the primary disease site.
  Disease progression was defined using either the RECIST or Pet criteria. Using the RECIST criteria disease progression is defined as a more than 25% tumor increase by volume and/ or presence of a new lesion. Using the Pet criteria disease progression is defined as an increase in PET activity as compared to the scan used in the planning of the treatment; any subsequent increase in SUVmax was defined as local progression.
Time Frame: up to 3 years
Measure: Number; unit: participants
Groups:
- Stereotactic Radiosurgery: patients w/ pancreas Cancer receiving Stereotactic Radiosurgery and Gemcitabine
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 20
participants | 15 [0 to 24 months]
Statistical Analysis 1: Comparison: Stereotactic Radiosurgery; Test type: Superiority or Other; proportion = .75

2. Secondary Outcome: Median Overall Survival Time
Description: The survival time for each patient is measured as the number of months from randomization until the time of death from any cause. The median survival time is computed using Kaplan Meier curves.
Time Frame: up to 3 years
Measure: Median (Full Range); unit: months
Groups:
- Stereotactic Body Radiotherapy: single fraction 25 Gy dose Stereotactic Body Radiotherapy on Trilogy Linear Accelerator, followed by weekly Gemcitabine
  Stereotactic Body Radiotherapy: Stereotactic Body Radiotherapy will be performed using Trilogy Linear Accelerator
  Gemcitabine: Weekly Gemcitabine will be administered at 1000mg/m2 over 100 minutes
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 20
months | 11.8 [7 to 25.1]

ADVERSE EVENTS:
Time Frame: following SBRT, follow-up at 4-6 weeks, then every 3 months in year 1 and 4 months year 2.
Groups:
- SBRT With Gem: patient with locally advanced pancreas cancer receiving Gem + SBRT
Arm/Group | SBRT With Gem
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 6/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT With Gem (N=20)
Perforation (Gastrointestinal disorders) | 1 (1) — duodenal perforation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT With Gem (N=20)
pain (Gastrointestinal disorders) | 1 (1) — pain
vomiting (Gastrointestinal disorders) | 2 (2)
ulcer (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes